CLINICAL TRIAL: NCT02550847
Title: Evaluation of Prognosis With Integrated MRI/PET in Patients With Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201407052MINC
Record Dates: First submitted 2015-09-08; First posted 2015-09-16 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Pancreatic Cancer
Keywords: MR/PET; pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: The imaging biomarkers determined by MR-PET — The aim of this study was to evaluate MR/PET with both functional and molecular imaging on the prediction of prognosis in patients with suspected pancreatic cancer.

SUMMARY:
The aim of this study was to evaluate MR/PET with both functional and molecular imaging on the prediction of prognosis in patients with suspected pancreatic cancer.

DETAILED DESCRIPTION:
The results of MR/PET will be compared prospectively to dedicated MDCT or MR imaging, pathologic results, and clinical outcomes to assess the value of MR/PET in pancreatic cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as pancreatic cancer
2. Between 20~90 years old
3. ECOG 0-2
4. Normal renal function
5. Measurable tumor size (>1cm)

Exclusion Criteria:

1. Contraindication for MRI exam
2. Claustrophobia
3. Renal insufficiency
4. Other malignancy
5. Pregnancy and lactating women

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include 100 consecutive patients (around 100 newly diagnosed patients per year at NTUH) presenting with suspect pancreatic cancer for treatment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-04 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
The tumor recurrence rate after operation at 6 months | 6 months

SECONDARY OUTCOMES:
The overall survival after operation at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ting-Fang Shih, MD, Principal Investigator — Department of Medical Imaging, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan